CLINICAL TRIAL: NCT03044704
Title: Influence of Haemodynamic and Geometric Factors on the Onset and Progression of Atherosclerosis
Brief Title: Haemodynamic and Geometric Factors in Atherosclerosis
Acronym: ANGLE
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Peter Marschang, Ao. Univ.Prof.Dr., Medical University Innsbruck
Other Study IDs: AN2016-0189 366/4.4
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective-observational, explorative single-centre cohort study aimed to examine the influence of hemodynamic and geometric parameters on the progression of atherosclerotic alterations in peripheral vessels (carotids, femoral artery). Atherosclerotic alterations (IMT, plaque volume) will be measured with a ultrasound (IMT measurements and 3D quantitative plaque volumetry) and magnetic resonance imaging (MRI). Geometric parameters (e.g. carotid/femoral bifurcation angle, carotid/femoral bifurcation area) are assessed with magnetic resonance imaging (MRI) and also 3D ultrasonography.

A total of 100 patients with an asymmetrical plaque distribution in carotid and femoral arteries will be tested. Only patients who are already enrolled in the "Correlation of Artherosclerotic Plaque Volume and Intima Media Thickness With Soluble P-selectin" (NCT01895725) and who are tested prior for an asymmetrical plaque distribution will be included in this study. MRI will be performed once whereas ultrasound imaging will be be repeated once per year (up to five times) to assess changes in these parameters over time. Also plasma samples will be collected once yearly and tested for traditional and novel cardiovascular risk factors.

The primary endpoint of the planned study will be the correlation between geometrical and hemodynamic parameters as stated above and the progression of atherosclerosis as measured by plaque volume and IMT in the carotid and femoral arteries, respectively.

Secondary endpoints will include the correlation of geometrical and hemodynamic parameters with established (hypertension, smoking, diabetes, dyslipidemia) and novel risk factors (hsCRP, P-selectin, cholesteryl ester transfer protein (CETP), intercellular adhesion molecule-1 (ICAM-1), CETP TaqIb polymorphism), with cardiovascular event rate, plaque localization, plaque morphology and the additional predictive value of geometrical parameters compared to an established risk score (SCORE card).

ELIGIBILITY:
Inclusion Criteria:

* asymmetrical (side difference) plaque distribution in carotids/femoral arteries which was tested in at least two prior 3D-ultrasound examinations (absolute side difference in carotid arteries ≥ 30 mm3 or in femoral arteries ≥50 mm3 and relative side difference in carotid arteries/femoral arteries ≥50% )

Exclusion Criteria:

* actual pregnancy, lactation period, chronic renal insufficiency (GFR<20ml/min)

Ages: 30 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Only patients who are already enrolled in the "Correlation of Artherosclerotic Plaque Volume and Intima Media Thickness With Soluble P-selectin" (NCT01895725) and who are tested prior for an asymmetrical plaque distribution will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between geometrical and hemodynamic parameters and the progression of atherosclerosis | up to 1 year
  Haemodynamic/geometric parameters will be assessed with MRI and 3D-US. This includes carotid/femoral bifurcation angle, common carotid/femoral area, carotid/femoral bifurcation area, internal and external carotid area, femoral superficial artery area and carotid/femoral bifurcation length. Progression of atherosclerosis will be measured via 3D-US by plaque volume and IMT in the carotid and femoral arteries, respectively.

SECONDARY OUTCOMES:
Correlation of geometrical and hemodynamic parameters with established and novel risk factors. | up to 1 year
  Secondary endpoint will include the correlation of geometrical and hemodynamic parameters with established (hypertension, smoking, diabetes, dyslipidemia) and novel risk factors (hsCRP, P-selectin, cholesteryl ester transfer protein (CETP), intercellular adhesion molecule-1 (ICAM-1), CETP TaqIb polymorphism), with cardiovascular event rate, plaque localization, plaque morphology and the additional predictive value of geometrical risk constellations compared to an established risk score (SCORE card).
Correlation of geometrical and hemodynamic parameters with cardiovascular event rate | 1 year
  Secondary endpoint will include the correlation of geometrical and hemodynamic parameters with the cardiovascular event rate (MACE-rate, coronary/ femoral surgery/intervention)
Correlation of geometrical and hemodynamic parameters with plaque morphology | up to 1 year
  Secondary endpoint will include the correlation of geometrical and hemodynamic parameters with the plaque morphology (gray-scale median, Gray-Weale scores, plaque surface state)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Marschang, Prof., MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schreinlechner M, Noflatscher M, Kremser C, Steiger R, Gromer J, Theurl M, Kirchmair R, Mayr A, Marschang P. A Large Bifurcation Angle Is Strongly Associated With Increased Plaque Volume and Plaque Progression. JACC Cardiovasc Imaging. 2019 Oct;12(10):2087-2088. doi: 10.1016/j.jcmg.2019.05.006. Epub 2019 Jun 12. No abstract available. PMID 31202757